CLINICAL TRIAL: NCT06300229
Title: Novel Approach for Oligospermia (NAPO): A Randomized Controlled Trial
Brief Title: NAPO - Novel Approach for Oligospermia
Acronym: NAPO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Head of Research Department Endocrinology, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-508325-27-00
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Denosumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Active Comparator): Subcutaneous injection with 60 mg Denosumab once
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Subcutaneous injection with NaCl once
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injection with 60 mg Denosumab once
  Other Names: Prolia
  Arms: Denosumab
Drug: sodium chloride — Subcutaneous injection with NaCl once
  Other Names: sodium chloride (NaCl)
  Arms: Placebo

SUMMARY:
This randomized controlled trial aims to assess whether treatment with denosumab can improve semen quality in infertile men selected by serum anti-mullerian hormone (AMH) as a positive predictive biomarker, and with severely impaired semen quality (concentrations between 0.01 million/mL to 2 million/mL).

DETAILED DESCRIPTION:
Infertility is a common problem globally and impaired semen quality is responsible for up to 40% of all cases. Despite the high prevalence there are currently only very limited treatment options to improve semen quality for infertile men. Instead, almost all infertile couples are treated with inseminations or assisted reproductive techniques (ARTs) independently of the etiology of infertility. ARTs are very successful but expensive and associated with a significant treatment burden of the female partner due to the invasive methodology and the need for hormonal treatment often for several months.

RANKL is a ligand for the receptor activator of nuclear factor kappa beta (RANK), and their pathway plays a prominent role in the regulation of bone metabolism. The binding of RANKL to RANK on osteoclast precursors induces osteoclast maturation and activation, thereby stimulating bone resorption, and regulates cell cycle i.e., proliferation, differentiation, and apoptosis. Osteoprotegerin (OPG) is a secreted decoy receptor that controls RANKL-RANK interaction by binding RANKL and inhibits activation of RANK and preventing osteoclast differentiation and activation.

Denosumab, a drug used in millions of patients worldwide under trade names Prolia® and Xgeva®, inhibits the RANKL pathway and is used to treat osteoporosis and bone metastases. The drug's mechanism of action inhibits RANKL and thus inhibits bone resorption through reduced osteoclast activation. This reduces the loss of bone mineral density (BMD), which reduces the risk of bone loss and thereby the risk of fracture and osteoporosis. Denosumab has been shown in several clinical studies to be a safe and effective drug in both women and men and has been in clinical use in both sexes for many years. As Denosumab has a teratogenic effect, pharmacokinetic studies in both monkeys and healthy men were performed before approval of the drug as a treatment for osteoporosis in men. These studies showed that Denosumab concentration in semen does not pose a risk to the fetus during sexual intercourse with the pregnant woman and therefore is safe to use for the suggested infertility indication as there is no risk of fetal transmission.

In light of this, our research group has investigated the effect of denosumab in human testicular germ cell lines as well as in human testicular tissue ex vivo "hanging drop" cultures. Treatment with denosumab did in both cases increase the proliferation of the germinal cells, which is an indicator that denosumab treatment potential beneficial effect on sperm production by reducing apoptosis in the germ cells. This led to a pilot intervention study of 12 infertile men who were overall healthy and without comorbidities. The men were treated with a single-dose of 60 mg of denosumab subcutaneous (s.c.). The study showed that the response to RANKL inhibition was either bad or highly beneficial. This was an interesting finding and indicates that only a fraction of infertile men should be offered denosumab treatment and this fraction of beneficial responders should ideally be identified based on an easily accessible biomarker before initiation of treatment. On this knowledge, a randomized controlled trial, "First In Treating Male Infertility" (FITMI), is being conducted to explore whether treatment with denosumab can improve semen quality in infertile men who are selected by serum AMH, but already have a sperm concentration that is at least 2 million/mL. This is an important study, but unfortunately, it leaves out a solution for those with sperm concentration under 2 million/mL, who are the most vulnerable in this regard. Therefore, there is a need for a randomized controlled trial that addresses the specific concerns of individuals with sperm concentrations below 2 million/mL to provide a valuable option in an otherwise hopeless situation.

NAPO is a single-center, sponsor-investigator-initiated, placebo-controlled, double-blinded randomized trial. Following successful completion of screening procedures, subjects will be randomized in a 2:1 fashion to receive either denosumab 60 mg s.c. or a placebo. The study will be carried out at the Division of Translational Endocrinology, Copenhagen University Hospital, Herlev, Copenhagen, Denmark.

With the power to avoid a type II error set to 80% (1-β) at a two-sided 5% significance level, 42 men allocated 2:1 in each of the investigation arms are needed to detect a difference in sperm concentration of 100% between intervention and placebo group in the primary outcome. The primary analysis will be a covariance analysis in which day 80 measurements are analyzed, initially as crude values but also adjusted on baseline.

ELIGIBILITY:
Inclusion Criteria:

* Infertile men ≥ 18 years and < 60 years of age
* Sperm concentration ≤ 2 million pr. mL
* Serum AMH levels ≥28 pmol/L.
* The participants must have appropriate Danish or English language skills and give written informed consent.

Exclusion Criteria:

* Chronic diseases, defined as diagnosis where signs, symptoms, and treatment imply an expected long duration and lack of a cure, such as diabetes mellitus, metabolism disorders, osteoporosis, colitis, etc.
* Sperm concentration <0.01 million pr. mL
* Men with current or previous malignancies, or at potential risk of testicular cancer after baseline examination and ultrasound will be excluded.
* Men with hypocalcemia at baseline, defined as albumin corrected calcium < 2,17 mmol/L or total calcium < 2.14 mmol/L
* Serum vitamin D (25OHD) levels < 25 nmol/L
* estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1,73 m2
* Insufficient dental status
* Vasectomy
* Hypersensitivity to latex, Denosumab, or to any of the excipients (acetic acid, sodium hydroxide, Sorbitol (E420), Polysorbate 20) will be excluded.
* Serum FSH <3 IU/L
* Testis size > 17 mL
* BMI ≥ 35 kg/m2

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
The difference in sperm concentration (million pr. mL) on day 80 | Day 80 and day 83 after inclusion
  Semen analysis - The average concentration of two semen samples delivered on day 80 and day 83 after inclusion is used.

SECONDARY OUTCOMES:
The difference in semen quality (total sperm count, motile sperm, progressive motile sperm and morphologically normal sperm) between baseline and two semen samples delivered at day 80 and day 83 after inclusion | Day 80 and day 83 after inclusion
  Semen analysis
The change/differences in number of pregnancies achieved before day 180 | Day 180 after inclusion
  Survey
The difference in the number of miscarriages throughout the trial before day 180 | Day 450 after inclusion]
  Survey
The change/difference in serum levels of follicle stimulating hormone (FSH) on day 80 | Day 80 after inclusion
  Serum sample
The change/difference in serum levels of reproductive hormone luteinizing hormone (LH) on day 80 | Day 80 after inclusion
  Serum sample
The change/difference in serum levels of reproductive hormone AMH on day 80 | Day 80 after inclusion
  Serum sample
The change/difference in serum levels of reproductive hormone Inhibin B on day 80 | Day 80 after inclusion
  Serum sample

OTHER OUTCOMES:
The change/difference in CatSper expression on day 80 | Day 80 after inclusion
  Seminal fluid
The change/difference in RANKL expression on day 80 | Day 80 after inclusion
  Seminal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kafai Yahyavi, MD, Principal Investigator — Division of Translational Endocrinology, Herlev, Copenhagen
Locations (1):
- Division of Translational Endocrinology, Department of Endocrinology and Internal Medicine, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huynh T, Mollard R, Trounson A. Selected genetic factors associated with male infertility. Hum Reprod Update. 2002 Mar-Apr;8(2):183-98. doi: 10.1093/humupd/8.2.183. PMID 12099633
- [Background] Krausz C. Male infertility: pathogenesis and clinical diagnosis. Best Pract Res Clin Endocrinol Metab. 2011 Apr;25(2):271-85. doi: 10.1016/j.beem.2010.08.006. PMID 21397198
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Buck Louis GM, Toppari J, Andersson AM, Eisenberg ML, Jensen TK, Jorgensen N, Swan SH, Sapra KJ, Ziebe S, Priskorn L, Juul A. Male Reproductive Disorders and Fertility Trends: Influences of Environment and Genetic Susceptibility. Physiol Rev. 2016 Jan;96(1):55-97. doi: 10.1152/physrev.00017.2015. PMID 26582516
- [Background] Blomberg Jensen M, Lawaetz JG, Petersen JH, Juul A, Jorgensen N. Effects of Vitamin D Supplementation on Semen Quality, Reproductive Hormones, and Live Birth Rate: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Mar 1;103(3):870-881. doi: 10.1210/jc.2017-01656. PMID 29126319
- [Background] Bollehuus Hansen L, Kaludjerovic J, Nielsen JE, Rehfeld A, Poulsen NN, Ide N, Skakkebaek NE, Frederiksen H, Juul A, Lanske B, Blomberg Jensen M. Influence of FGF23 and Klotho on male reproduction: Systemic vs direct effects. FASEB J. 2020 Sep;34(9):12436-12449. doi: 10.1096/fj.202000061RR. Epub 2020 Jul 30. PMID 32729975
- [Background] Juel Mortensen L, Lorenzen M, Jorgensen N, Andersson AM, Nielsen JE, Petersen LI, Lanske B, Juul A, Hansen JB, Blomberg Jensen M. Possible link between FSH and RANKL release from adipocytes in men with impaired gonadal function including Klinefelter syndrome. Bone. 2019 Jun;123:103-114. doi: 10.1016/j.bone.2019.03.022. Epub 2019 Mar 23. PMID 30914274
- [Background] Blomberg Jensen M. Vitamin D and male reproduction. Nat Rev Endocrinol. 2014 Mar;10(3):175-86. doi: 10.1038/nrendo.2013.262. Epub 2014 Jan 14. PMID 24419359
- [Background] Kearns AE, Khosla S, Kostenuik PJ. Receptor activator of nuclear factor kappaB ligand and osteoprotegerin regulation of bone remodeling in health and disease. Endocr Rev. 2008 Apr;29(2):155-92. doi: 10.1210/er.2007-0014. Epub 2007 Dec 5. PMID 18057140
- [Background] Lacey DL, Timms E, Tan HL, Kelley MJ, Dunstan CR, Burgess T, Elliott R, Colombero A, Elliott G, Scully S, Hsu H, Sullivan J, Hawkins N, Davy E, Capparelli C, Eli A, Qian YX, Kaufman S, Sarosi I, Shalhoub V, Senaldi G, Guo J, Delaney J, Boyle WJ. Osteoprotegerin ligand is a cytokine that regulates osteoclast differentiation and activation. Cell. 1998 Apr 17;93(2):165-76. doi: 10.1016/s0092-8674(00)81569-x. PMID 9568710
- [Background] Simonet WS, Lacey DL, Dunstan CR, Kelley M, Chang MS, Luthy R, Nguyen HQ, Wooden S, Bennett L, Boone T, Shimamoto G, DeRose M, Elliott R, Colombero A, Tan HL, Trail G, Sullivan J, Davy E, Bucay N, Renshaw-Gegg L, Hughes TM, Hill D, Pattison W, Campbell P, Sander S, Van G, Tarpley J, Derby P, Lee R, Boyle WJ. Osteoprotegerin: a novel secreted protein involved in the regulation of bone density. Cell. 1997 Apr 18;89(2):309-19. doi: 10.1016/s0092-8674(00)80209-3. PMID 9108485
- [Background] Khosla S. Minireview: the OPG/RANKL/RANK system. Endocrinology. 2001 Dec;142(12):5050-5. doi: 10.1210/endo.142.12.8536. PMID 11713196
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Makras P, Polyzos SA, Papatheodorou A, Kokkoris P, Chatzifotiadis D, Anastasilakis AD. Parathyroid hormone changes following denosumab treatment in postmenopausal osteoporosis. Clin Endocrinol (Oxf). 2013 Oct;79(4):499-503. doi: 10.1111/cen.12188. Epub 2013 Apr 1. PMID 23452098
- [Background] Schwarz P, Rasmussen AQ, Kvist TM, Andersen UB, Jorgensen NR. Paget's disease of the bone after treatment with Denosumab: a case report. Bone. 2012 May;50(5):1023-5. doi: 10.1016/j.bone.2012.01.020. PMID 22586699
- [Background] Polyzos SA, Singhellakis PN, Naot D, Adamidou F, Malandrinou FC, Anastasilakis AD, Polymerou V, Kita M. Denosumab treatment for juvenile Paget's disease: results from two adult patients with osteoprotegerin deficiency ("Balkan" mutation in the TNFRSF11B gene). J Clin Endocrinol Metab. 2014 Mar;99(3):703-7. doi: 10.1210/jc.2013-3762. Epub 2014 Jan 16. PMID 24433001
- [Background] Papapoulos S, Chapurlat R, Libanati C, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Man Z, Mellstrom D, Radominski SC, Reginster JY, Resch H, Roman Ivorra JA, Roux C, Vittinghoff E, Austin M, Daizadeh N, Bradley MN, Grauer A, Cummings SR, Bone HG. Five years of denosumab exposure in women with postmenopausal osteoporosis: results from the first two years of the FREEDOM extension. J Bone Miner Res. 2012 Mar;27(3):694-701. doi: 10.1002/jbmr.1479. PMID 22113951
- [Background] Boonen S, Adachi JD, Man Z, Cummings SR, Lippuner K, Torring O, Gallagher JC, Farrerons J, Wang A, Franchimont N, San Martin J, Grauer A, McClung M. Treatment with denosumab reduces the incidence of new vertebral and hip fractures in postmenopausal women at high risk. J Clin Endocrinol Metab. 2011 Jun;96(6):1727-36. doi: 10.1210/jc.2010-2784. Epub 2011 Mar 16. PMID 21411557
- [Background] Sohn W, Lee E, Kankam MK, Egbuna O, Moffat G, Bussiere J, Padhi D, Ng E, Kumar S, Slatter JG. An open-label study in healthy men to evaluate the risk of seminal fluid transmission of denosumab to pregnant partners. Br J Clin Pharmacol. 2016 Feb;81(2):362-9. doi: 10.1111/bcp.12798. Epub 2015 Dec 5. PMID 26447647
- [Background] Bussiere JL, Pyrah I, Boyce R, Branstetter D, Loomis M, Andrews-Cleavenger D, Farman C, Elliott G, Chellman G. Reproductive toxicity of denosumab in cynomolgus monkeys. Reprod Toxicol. 2013 Dec;42:27-40. doi: 10.1016/j.reprotox.2013.07.018. Epub 2013 Jul 22. PMID 23886817
- [Background] Uhland AM, Kwiecinski GG, DeLuca HF. Normalization of serum calcium restores fertility in vitamin D-deficient male rats. J Nutr. 1992 Jun;122(6):1338-44. doi: 10.1093/jn/122.6.1338. PMID 1588451
- [Background] Kwiecinski GG, Petrie GI, DeLuca HF. Vitamin D is necessary for reproductive functions of the male rat. J Nutr. 1989 May;119(5):741-4. doi: 10.1093/jn/119.5.741. PMID 2723823
- [Background] Jorgensen A, Blomberg Jensen M, Nielsen JE, Juul A, Rajpert-De Meyts E. Influence of vitamin D on cisplatin sensitivity in testicular germ cell cancer-derived cell lines and in a NTera2 xenograft model. J Steroid Biochem Mol Biol. 2013 Jul;136:238-46. doi: 10.1016/j.jsbmb.2012.10.008. Epub 2012 Oct 23. PMID 23098692
- [Background] Blomberg Jensen M, Jorgensen A, Nielsen JE, Steinmeyer A, Leffers H, Juul A, Rajpert-De Meyts E. Vitamin D metabolism and effects on pluripotency genes and cell differentiation in testicular germ cell tumors in vitro and in vivo. Neoplasia. 2012 Oct;14(10):952-63. doi: 10.1593/neo.121164. PMID 23097629
- [Background] Blomberg Jensen M, Lieben L, Nielsen JE, Willems A, Jorgensen A, Juul A, Toppari J, Carmeliet G, Rajpert-De Meyts E. Characterization of the testicular, epididymal and endocrine phenotypes in the Leuven Vdr-deficient mouse model: targeting estrogen signalling. Mol Cell Endocrinol. 2013 Sep 5;377(1-2):93-102. doi: 10.1016/j.mce.2013.06.036. Epub 2013 Jul 11. PMID 23850520
- [Background] Blomberg Jensen M, Andreassen CH, Jorgensen A, Nielsen JE, Juel Mortensen L, Boisen IM, Schwarz P, Toppari J, Baron R, Lanske B, Juul A. RANKL regulates male reproductive function. Nat Commun. 2021 Apr 23;12(1):2450. doi: 10.1038/s41467-021-22734-8. PMID 33893301
- [Background] Adler RA, Gill RS. Clinical utility of denosumab for treatment of bone loss in men and women. Clin Interv Aging. 2011;6:119-24. doi: 10.2147/CIA.S14565. Epub 2011 May 24. PMID 21753866
- [Background] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Background] Lunenfeld B, Van Steirteghem A; Bertarelli Foundation. Infertility in the third millennium: implications for the individual, family and society: condensed meeting report from the Bertarelli Foundation's second global conference. Hum Reprod Update. 2004 Jul-Aug;10(4):317-26. doi: 10.1093/humupd/dmh028. Epub 2004 Jun 10. PMID 15192057
- [Background] Yahyavi SK, Holt R, Knudsen NK, Andreassen CH, Sejling C, Meddis A, Kjaer SK, Schwarz P, Jensen JB, Torp-Pedersen C, Juul A, Selmer C, Blomberg Jensen M. Cancer risk in patients treated with denosumab compared with alendronate: A population-based cohort study. Bone. 2024 May;182:117053. doi: 10.1016/j.bone.2024.117053. Epub 2024 Feb 21. PMID 38395247
- [Background] Yahyavi SK, Holt R, Juel Mortensen L, Petersen JH, Jorgensen N, Juul A, Blomberg Jensen M. Effect of a single-dose denosumab on semen quality in infertile men (the FITMI study): study protocol for a randomized controlled trial. Trials. 2022 Jun 22;23(1):525. doi: 10.1186/s13063-022-06478-4. PMID 35733213
- [Derived] Yahyavi SK, Jorsal MJ, Holt R, Nohr B, Blomberg Jensen M. Novel approach for oligospermia (NAPO) - Protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2024 Aug 22;41:101352. doi: 10.1016/j.conctc.2024.101352. eCollection 2024 Oct. PMID 39280787